CLINICAL TRIAL: NCT03120754
Title: Clinical Study of Abdominal Drainage in Laparoscopic Common Bile Duct Exploration With Primary Closure
Brief Title: Study of Abdominal Drainage in LCBDE+PC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhongshan Hospital Xiamen University (Other)
Responsible Party: Principal Investigator, Jianyin Zhou, Chief physician, Zhongshan Hospital Xiamen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 011314
Record Dates: First submitted 2017-04-07; First posted 2017-04-19 (Actual); Last update posted 2017-04-19 (Actual); Status verified 2017-03

CONDITIONS: Enhanced Recovery After Surgery
Keywords: ERAS; Peritoneal drainage; Primary Closure

STUDY DESIGN:
Intervention Model Description: SPSS statistical analysis system by the deputy director of our department physician, accepted treatment of 80 subjects (test group and control group) randomly arranged, which lists the serial number from 1 to 80 corresponding to the treatment assignment. In the experiment, 1 patients were divided into the exper
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Placement of peritoneal drainage
  Interventions: Procedure: Place the peritoneal drainage
- Control group (Active Comparator): No peritoneal drainage
  Interventions: Procedure: No peritoneal drainage

INTERVENTIONS:
Procedure: Place the peritoneal drainage — In the experimental group, the abdominal drainage was not placed
  Arms: Experimental Group
Procedure: No peritoneal drainage — Intraoperative placement of peritoneal drainage as control group.
  Arms: Control group

SUMMARY:
Common bile duct stones in clinical manifestations of biliary colic, obstructive jaundice, cholangitis, pancreatitis and other symptoms. At present, thanks to the rapid development of minimally invasive surgery and the concept of ERAS, laparoscopic common bile duct incision and primary suture has been gradually used as a routine surgical approach in clinical application. However, whether or not to place the abdominal drainage tube after surgery, so far has not yet reached a consensus. Therefore, this study focuses on the clinical advantages of LCBDE+PC placed abdominal drainage.

DETAILED DESCRIPTION:
On the basis of the analysis of 7 cases were selected by laparoscopic treatment of cholecystolithiasis complicated with choledocholithiasis bile duct suture in patients with a clinical data of our hospital were prospectively divided into peritoneal drainage group of 40 cases, no abdominal drainage group of 40 cases, compared two groups of operation time, hospitalization time and cost, operation cost, operation bleeding and postoperative bilirubin recovery, complication and return to hospital again and so on, and to explore the clinical significance of indwelling drainage tube.

ELIGIBILITY:
Inclusion Criteria:

* cholecystocholedocholithiasis or simple choledocholithiasis, no intrahepatic bile duct stones, bile duct diameter greater than 8 mm;
* no acute suppurative cholangitis or severe acute biliary pancreatitis;
* all patients were treated with internal medicine before operation, such as anti inflammation, liver protection, correction of anemia, hypoproteinemia, disturbance of electrolyte and acid-base imbalance;
* there was no obvious stenosis of common bile duct;
* aged from 18 to 80 years;
* BMI<30 kg / m2;
* American Society of anesthesiologists (ASA) anesthesia risk rating of 1 or 2.

Exclusion Criteria:

* severe anemia or thrombocytopenia in patients with 50*109/L, PT is greater than 15s and can not correct the coagulation disorders;
* severe heart and lung complications can not tolerate pneumoperitoneum and other laparoscopic surgery contraindications;
* IgG4 associated cholangitis and other immune system diseases;
* there is a serious systemic disease. The patients with the following conditions:

  * there was inflammatory stenosis or Oddi sphincter hyperemia and edema at the lower end of the common bile duct;
  * in acute inflammation in patients with obstructive jaundice, such patients have biliary dilatation, the bile duct wall edema obviously and easily with bile duct opening at the lower end of the inflammatory edema, biliary high pressure, suture of bile duct after prone to bile leakage;
  * the presence of severe cholangitis requiring emergency biliary drainage;
  * it is difficult to get a combination of intrahepatic bile duct stones and choledochoscopy;
  * Mirizzi syndrome type II-IV.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-03-24 (Actual); Primary Completion 2018-07-30 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Hospital stay | 3 days
  length of patient stay.

SECONDARY OUTCOMES:
Postoperative pain | 24 and 48hours
  Observation on pain after operation in the two groups, were evaluated according to the standard for evaluation of VAS pain score.

OTHER OUTCOMES:
Complication | 6 month
  The postoperative complications were compared, such as bile leakage, abdominal infection and so on.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of hepatobiliary and pancreatic surgery; Zhongshan Hospital Affiliated to Xiamen University, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: Undecided